CLINICAL TRIAL: NCT05871333
Title: Effect of Losartan on the Incidence and Severity of Chemotherapy-Induced Mucositis in Gastrointestinal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amira Yousry, Clinical Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Losartan, Mucositis
Record Dates: First submitted 2023-03-15; First posted 2023-05-23 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Chemotherapy; Colorectal Cancer; Intestinal Mucositis; Oral Mucositis
Keywords: Losartan; Colorectal Cancer; Chemotherapy-Induced Mucositis
MeSH Terms: conditions — Colorectal Neoplasms; Stomatitis | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: Group I: Patients will receive only their standard therapy for 4 months. Group II: will receive the studied drug orally in addition to their standard therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Patients will receive FOLFOX-6 regimen consisted of 2-hour infusion of oxaliplatin (100 mg/m2) and 2-hour infusion of leucovorin (400 mg/m2) on Day 1, followed by 5-fluorouracil (5-FU) bolus (400 mg/ m2) on Day 1 and 46-hour infusion (2.4 g/m2) with cycle repeated every 2 weeks over range of 20-24 weeks depending on patients disease state.
- standard of care + Losartan (Experimental): Patients will receive FOLFOX-6 regimen consisted of 2-hour infusion of oxaliplatin (100 mg/m2) and 2-hour infusion of leucovorin (400 mg/m2) on Day 1, followed by 5-fluorouracil (5-FU) bolus (400 mg/ m2) on Day 1 and 46-hour infusion (2.4 g/ m2) with cycle repeated every 2 weeks over range of 20-24 weeks depending on patients disease state. In addition to Losartan 50 mg/day orally for 4 months.
  Interventions: Drug: Losartan 50mg Tab

INTERVENTIONS:
Drug: Losartan 50mg Tab — Losartan 50 mg oral tablets
  Other Names: Angiotension receptor blockers
  Arms: standard of care + Losartan

SUMMARY:
Mucositis is a common and clinically significant side effect of both anticancer chemotherapy and radiation therapy that can affect any portion of the gastrointestinal tract. Not only associated with an adverse symptom profile, but also it may limit patients' ability to tolerate treatment if not adequately prevented and managed. Moreover, it may be associated with secondary local and systemic infection and poor health outcomes, and generates additional use of healthcare resources resulting in additional costs.

Based on study of 38 patients of mean age sixty-one years old diagnosed with colorectal carcinoma were included to evaluate gastrointestinal adverse effect with different schedules of FOLFOX. Incidence of oral mucositis with FOLFOX-4 Is 76%, FOLFOX-6 is 62%, mFOLFOX-6 is 79% and FOLFOX-7 is 93%

Chemotherapy-induced mucositis is commonly described as a five-phase sequence:

initiation (0-2 days),upregulation and activation of messengers (2-3 days), signal amplification (2-5 days), ulceration with inflammation (5-14 days) and healing (14-21 days)

According to the model introduced by some studies the primary inducer involved in unleashing mucosal injury upon chemotherapy is the production of reactive oxygen species (ROS), leading to tissue inflammation and mucositis induction.

Inflammatory signaling pathways are upregulated during high reactive oxygen species states which further contribute to cytotoxicity. leading to the third step in the oral mucositis pathway. In this inflammatory phase, cytokines including Tissue Necrosis Factor alpha (TNF-α), prostaglandins, Nuclear factor Kappa β (NF-кβ), and interleukin (IL) 1β are released.

The cytotoxic effects of chemotherapy, inflammation, and reactive oxygen species-mediated DNA damage result in gradual apoptosis of mucosal epithelial cells. Ulcerative sites become relatively neutropenic which predisposes them to bacterial and yeast infections. These bacterial toxins further simulate the underlying inflammatory state through release of additional cytokines.

It is necessary to emphasize that oral mucositis is frequently documented only in its advanced phases owing to the requirements for clinical therapy and assistance. Therefore, the search for new active ingredients that could be used in the prevention (and even treatment) of oral and intestinal mucositis is of utmost importance.

DETAILED DESCRIPTION:
in this study Losartan, a AT1 angiotensin 2 receptor blockers (ARB), used clinically for antihypertensive purposes, has anti-inflammatory effects widely described in the literature.

Losartan has been shown to reduce pro-inflammatory cytokines, such as TNF-α, IL-1β, IL-6, and the activation of nuclear transcription factor (NF-κB), in addition to an antioxidant effect in different inflammatory diseases as neuropathic pain in patients with paclitaxel- induced peripheral neuropathy.

Studies have already shown that angiotensin 2 pathway modulators have a protective effect on oral and intestinal mucositis in rats.

Patients meeting the study inclusion criteria will be educated firmly about the disease details and all information about the drug, then will be assigned to one of two groups, the control group or the intervention group.

The two groups will undergo baseline evaluation at the beginning of the study including Demographic data collection: Age, gender, weight, height, BSA, Risk factors related to mucositis, Medical history and Comorbidities reporting as HTN, DM and others, Vital signsas Blood pressure and pulse recording, Social history and Smoking status and Clinical assessment for confirmation of absence of mucositis and examination of oral mucous membrane and gut functions (bowel habits) Weekly for assessment of the following: occurrence and severity of OM and IM, Pain assessment will be done using the NRS score and through patient interview, occurrence and severity of dysphagia and Need for supportive management e.g. Painkillers and anti-diarrhea.

Every cycle for the need for hospitalization due to oral or intestinal symptoms or any unplanned chemotherapy breaks due to oral or intestinal toxicity in both groups.

In between cycles via phones for any side effects encountered by patients in both groups due to the administered drug (Losartan). Patients will be given a side effects reporting card for follow up if any side effect occurred during treatment. And Quality of Life assessment by Functional Assessment of Cancer Therapy- General (FACT-G).

By the end of cycle 8, all patients in both groups will be reassessed for all laboratory and clinical evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years old or more.
2. Patients diagnosed with gastrointestinal cancer eligible for chemotherapy
3. Eastern Cooperative Oncology Group (ECOG) performance ≤ 2.
4. Platelet count more than 100 × 10^9/L.
5. Absolute neutrophil count: greater than 1.5 × 10^9/L.
6. Aspartate aminotransferase level up to 2.5 times the upper limit normal.
7. Serum bilirubin level not more than 1.5 times the institutional upper limit normal.
8. Serum creatinine levels up to 1.5 mg% and 1.4 mg% for males and females respectively.

Exclusion Criteria:

1. Currently taking an angiotensin converting enzyme inhibitor (ACEi) or Angiotensin receptor blocker (ARB)
2. Prior reaction or intolerance to an ARB or ACE inhibitor, including but not limited to angioedema.
3. Pregnant or breastfeeding women.
4. Females in child bearing age not currently taking a protocol allowed version of contraception: intrauterine device, Depo-formulation of hormonal contraception.
5. Patient reported history or electronic medical record history of kidney disease, defined as:

   Any history of dialysis. History of chronic kidney disease stage IV. Estimated Glomerular Filtration Rate (eGFR) of < 30ml/min/1.73 m2 Other Kidney disease that in the opinion of investigator, would affect Losartan Clearance.
6. Patient reported dehydration and significantly decreased urine output in the past 72 hours.
7. Most recent systolic blood pressure prior to enrollment <110 mmHg.
8. Current participation in any other clinical investigation.
9. Currently taking any drug contraindicated with Losartan administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-17 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Occurrence of oral mucositis | monthly for 6 months
  Assessment the occurrence of oral mucositis by physical examination of oral cavity
change in Severtity of Oral Mucositis | monthly for 6 months
  Assessment of the severity of oral mucositis using the national cancer institute common
change in severity of intestinal mucositis | monthly for 6 months
  assessment of the severity of oral mucositis using the national cancer institute terminology criteria version 5.0

SECONDARY OUTCOMES:
Evaluation of cancer control by Ultrasound | at Baseline and at week 24 ( end of study)
  Disease control will be assessed by US
Quality of life questionnaire | monthy for 6 months
  Adverse events encountered by patients in both groups, need for hospitalization due to oral and/or intestinal symptoms and unplanned chemotherapy breaks due to oral and/or intestinal toxicity will be recorded on weekly bases.
Laboratory evaluation of TNF-α level | baseline and at week 16
  Change in Tumor necrosis factor-a (TNF-α).
Laboratory evaluation of Interleukin-1β level | Baseline and at week 16
  Change in Interleukin-1β.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Y mohamed, Principal Investigator — Ain Shams University
Locations (1):
- Hospital, Cairo, Egypt